CLINICAL TRIAL: NCT01820013
Title: Management of Antenatal Pelvic Girdle Pain Study (MAPS): a Single Centre Blinded Randomized Trial Evaluating the Effectiveness of Two Pelvic Support Garments
Brief Title: Single Centre Blinded Randomized Controlled Trial Evaluating the Effectiveness of Two Pelvic Support Garments
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Jenny Freeman, Associate Professor (Reader) in Physiotherapy, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGP-LC12
Record Dates: First submitted 2013-03-15; First posted 2013-03-28 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Pelvic Pain; Symphysis Pubis Dysfunction
Keywords: Pelvic Girdle pain; Symphysis Pubis Dysfunction; Sacroiliac Joint; Sacroiliitis; Physiotherapy; Physical Therapy; Orthotic Devices
MeSH Terms: conditions — Pelvic Pain; Pelvic Girdle Pain; Sacroiliitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Customised Orthoses (Experimental): Customised Dynamic Elastomeric Fabric Orthoses (DEFO)
  Interventions: Device: Customised Dynamic Elastomeric fabric Orthoses
- Rigid 'off the shelf' pelvic support (Active Comparator): Serola Sacroiliac Belt.
  Interventions: Device: Serola Sacroiliac Belt

INTERVENTIONS:
Device: Customised Dynamic Elastomeric fabric Orthoses — Eligible participants will be measured and fitted with a customised Dynamic Elastomeric Fabric Orthoses. The participant may require a re-fitting of the garment as they progress through their pregnancy. Participants will also be issued with standardised advice on PGP management via an information leaflet from Association of Chartered Physiotherapists in Women's health website.
  Other Names: Customised Dynamic Elastomeric Fabric Orthoses (DEFO); Pelvic Support Garment
  Arms: Customised Orthoses
Device: Serola Sacroiliac Belt — Eligible participants will be measured and fitted with a Serola sacroiliac belt. Participants will also be issued with standardised advice on PGP management via an information leaflet from Association of Chartered Physiotherapists in Women's health website.
  Other Names: Rigid 'off the shelf' Pelvic Support Belt; Pelvic Support garment
  Arms: Rigid 'off the shelf' pelvic support

SUMMARY:
This blinded randomized comparative trial aims to determine the effectiveness of a customized Dynamic Elastomeric Fabric Orthoses (DEFO) compared to a standard pelvic belt in: a) reducing pregnancy-related pelvic girdle pain (PGP), b) optimizing activity levels in pregnant women with PGP, c) improving quality of life for pregnant women with PGP d) cost effectiveness.

DETAILED DESCRIPTION:
Pelvic girdle pain (PGP) occurs in an estimated 70% of pregnant women, of whom 25% have severe pain and 8% significant disability. Current methods of management, such as the use of rigid pelvic belts, are limited in their effectiveness. The Dynamic Elastomeric Fabric Orthoses (DEFO) has recently proven beneficial in managing PGP in athletes. There is a need to explore the potential use of DEFO for managing PGP during pregnancy. The primary aim of the study is to compare the effectiveness of a DEFO to a rigid 'off the shelf' pelvic support belt in terms of its effectiveness in reducing PGP during pregnancy. The secondary aims of the study are to compare the effectiveness of the DEFO to the rigid 'off the shelf' pelvic support belt in (a) optimizing activity levels in pregnant women with PGP, (b)improving quality of life for pregnant women with PGP. The relative cost effectiveness of these two interventions will also be compared.

ELIGIBILITY:
Inclusion Criteria:

women 20-36 weeks pregnant, who:

* report intermittent PGP (commenced or aggravated during pregnancy) which causes walking and/or stair climbing to be bothersome and
* are positive on at least 3 out of 7 pain provocation tests

Exclusion Criteria:

* recent history/signs or symptoms indicative of serious causes of pain that might be inflammatory, infective, traumatic, neoplastic, degenerative or metabolic, i.e. trauma, unexplained weight loss, history of cancer, steroid use, drug abuse, HIV infection, immunosuppressed state, neurological symptoms/signs such as: bowel, bladder, sensory, motor, reflex involvement (cauda equina, lumbar disk lesion, spinal stenosis,)
* fever
* systemically unwell
* obstetric complications
* pain that does not improve with rest/severe disabling pain
* history of chronic back or pelvic pain requiring surgery
* focal inflammatory signs/tenderness of spine (spondylolisthesis)
* known skin allergy to lycra
* >36 weeks pregnant (production of customized DEFO will take approximately 1 week)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Pain Levels | Baseline (pre intervention), 2 weekly intervals for potential of 20 weeks(pre-partum), 2 weekly intervals for 6 weeks (post-partum)
  Change in pain levels at 2 weekly intervals will be measured by a self report numerical rating scale.

SECONDARY OUTCOMES:
Change in Activity Levels | Baseline (pre intervention), 2 weekly intervals for potential of 20 weeks(pre-partum), 2 weekly intervals for 6 weeks (post-partum)
  Change in activity levels at 2 weekly intervals will be measured by a self report questionnaire.
Change in Quality of Life | Baseline (pre intervention), 2 weekly intervals for potential of 20 weeks(pre-partum), 2 weekly intervals for 6 weeks (post-partum)
  Change in Quality of life at two weekly intervals will be measured by two self report questionnaires:
  (i) Short Form 36 - Item Health Survey (Version 2) (ii) Euroqol (EQ-5D) Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cameron, Principal Investigator — University of Plymouth
Locations (2):
- United Kingdom (2):
  - Royal Cornwall Hospital, Truro, Cornwall
  - University of Plymouth, Plymouth, Devon

REFERENCES:
- [Background] Depledge J, McNair PJ, Keal-Smith C, Williams M. Management of symphysis pubis dysfunction during pregnancy using exercise and pelvic support belts. Phys Ther. 2005 Dec;85(12):1290-300. PMID 16305268
- [Background] Ekdahl L, Petersson K. Acupuncture treatment of pregnant women with low back and pelvic pain--an intervention study. Scand J Caring Sci. 2010 Mar;24(1):175-82. doi: 10.1111/j.1471-6712.2009.00704.x. Epub 2010 Jan 20. PMID 20102541
- [Background] Robinson HS, Mengshoel AM, Bjelland EK, Vollestad NK. Pelvic girdle pain, clinical tests and disability in late pregnancy. Man Ther. 2010 Jun;15(3):280-5. doi: 10.1016/j.math.2010.01.006. Epub 2010 Feb 8. PMID 20117040